CLINICAL TRIAL: NCT00513877
Title: An Open Label Phase II Multicentre Clinical Trial of Single Agent Bortezomib in Patients With Malignant Pleural Mesothelioma
Brief Title: Bortezomib in Treating Patients With Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-10 ICORG; ICORG-05-10; EUDRACT-2005-004420-39; EU-20748
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2013-01

CONDITIONS: Malignant Mesothelioma
Keywords: recurrent malignant mesothelioma; stage IA malignant mesothelioma; stage IB malignant mesothelioma; stage II malignant mesothelioma; stage III malignant mesothelioma; stage IV malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Bortezomib

ARMS (1):
- Bortezomib 1.6mg/m2 (Experimental)
  Interventions: Drug: bortezomib; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: bortezomib
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying the side effects of bortezomib and how well it works in treating patients with malignant pleural mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the clinical efficacy of bortezomib based on the evaluation of objective tumor response rate.

Secondary

* Assess additional clinical efficacy of bortezomib based on the evaluation of time to early disease progression and median overall 2-year survival rate.
* Assess safety and toxicity in these patients.
* Assess quality of life using the Lung Cancer Symptom Score.

OUTLINE: This is a multicenter study. Patients are stratified according to current treatment (first-line vs second-line)

Patients receive bortezomib IV on days 1, 8, 15, and 22. Treatment repeats every 5 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients exhibiting objective response or stable disease by week 20, may continue treatment at the discretion of the investigator until evidence of disease progression.

Quality of life is assessed periodically.

After completion of study treatment, patients are followed for up to 2 years.

PROJECTED ACCRUAL: 57 first-line setting and 54 second-line setting patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed malignant pleural mesothelioma
* Meets 1 of the following criteria for first-line or second-line chemotherapy:

  * Patients in the first-line setting must be unsuitable for, cannot access locally, or refuse combination chemotherapy
  * Patients in the second-line setting must be unsuitable for, cannot access locally, or refuse cytotoxic chemotherapy after failure of a first-line regimen

    * Second-line patients may not have received more than 1 prior line of antineoplastic treatment for this cancer
* Pleural effusions should be drained before treatment whenever possible

  * Talc or tetracycline pleurodesis may be used per standard practice for uncontrollable pleural effusions (recurrent despite regular drainage)

Exclusion criteria:

* Symptomatic or known brain or leptomeningeal metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* Hemoglobin ≥ 10 g/dL
* Neutrophil count ≥ 1,500 mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine clearance ≥ 30 mL/min
* AST and ALT < 3 times upper limit of normal
* Fertile patients must use effective contraception during study therapy

Exclusion criteria:

* Pregnant or breastfeeding
* History of prior malignant tumor within the past 3 years except for nonmelanoma skin tumor or carcinoma in situ of the cervix
* Patients suitably fit to receive a platinum doublet based chemotherapy (first-line only)
* Uncontrolled or severe cardiovascular disease including any of the following:

  * Myocardial infarction within the past 6 months
  * New York Heart Association class III or IV heart failure
  * Uncontrolled angina
  * Clinically significant pericardial disease
  * Cardiac amyloidosis
* Neuropathy ≥ grade 2 OR grade 1 with pain
* Serious medical (e.g., uncontrolled diabetes, hepatic disease, or infection) or psychiatric illness that would interfere with study participation
* Patients with known HIV or hepatitis B or C infection

PRIOR CONCURRENT THERAPY:

* No prior bortezomib
* No prior extensive radiation therapy, systemic chemotherapy, or other antineoplastic therapy within 4 weeks before enrollment
* No preplanned surgery or procedures that would interfere with the study
* More than 4 weeks since enrollment in another therapeutic clinical trial (i.e., received an experimental drug or used an experimental medical device)

  * Concurrent participation in non-treatment studies is allowed provided they do not interfere with participation in this study
* No concurrent experimental or antineoplastic agent other than bortezomib

  * Medications that may have antineoplastic activity, but are taken for other reasons than specific antineoplastic effect (e.g., megestrol [Megace®], cyclo-oxygenase-2 [COX-2] inhibitors, or bisphosphonates) are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate (complete response or partial response) as assessed by modified RECIST criteria | 28 days prior to baseline, at 10 weeks and at end of treatment
  The objective tumour response rate is a primary endpoint of the study. This will be a proportion of evaluable subjects who achieve a confirmed CR or PR per modified RECIST guidelines within four cycles (20 weeks) of treatment.

SECONDARY OUTCOMES:
Time to disease progression | Time to disease progression is measured from first treatment until the date of PD or death whichever is first reported. Subjects who did not progress or die will be censored at the day of their last tumour assessment.
Overall survival | Overall Survival is measured from the date of first treatment to the date of the subject's death. If the subject is alive or the vital status is unknown, the date of death will be censored at the date that the subject is last known to be alive.
Safety | The assessment of safety will be based mainly on the frequency of adverse events and on the number of laboratory values that fall outside of the pre-determined normal ranges.
Quality of life | Week 1, Week 10 and end of treatment
  Quality of life will be assessed using the Lung Cancer Symptom Score

CONTACTS AND LOCATIONS:
Overall Officials: Dean A. Fennell, MD, PhD, Principal Investigator — Centre for Cancer Research and Cell Biology at Queen's University Belfast
Locations (13):
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Ireland (7):
  - Cork University Hospital, Cork
  - Adelaide and Meath Hospital, Dublin Incorporating the National Children's Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Galway University Hospital, Galway
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands
- United Kingdom (4):
  - Saint Bartholomew's Hospital, London, England
  - Royal Marsden - Surrey, Sutton, England
  - Centre for Cancer Research and Cell Biology at Queen's University Belfast, Belfast, Northern Ireland
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland

REFERENCES:
- [Derived] Walter RFH, Sydow SR, Berg E, Kollmeier J, Christoph DC, Christoph S, Eberhardt WEE, Mairinger T, Wohlschlaeger J, Schmid KW, Mairinger FD. Bortezomib sensitivity is tissue dependent and high expression of the 20S proteasome precludes good response in malignant pleural mesothelioma. Cancer Manag Res. 2019 Sep 24;11:8711-8720. doi: 10.2147/CMAR.S194337. eCollection 2019. PMID 31576173